CLINICAL TRIAL: NCT04070222
Title: A Prospective Case-control Study of the Outcome and Influence Factors of Assisted Reproductive Therapy in Patients With Cesarean Scar Uterus.
Brief Title: The Outcome and Influence Factors of Assisted Reproductive Therapy in Patients With Cesarean Scar Uterus.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, MD, Sun Yat-sen University
Other Study IDs: newivf20190807
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Infertile Patients With Previous Live Birth
Keywords: Secondary infertility, cesarean section, post-cesarean section scar diverticulum , endometrial microflora, inflammatory markers, clinical pregnancy, live birth
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Natural labour group
  Interventions: Other: Hysteroscopy
- Cesarean scar group
  Interventions: Other: Hysteroscopy
- Cesarean with diverticulum (PCSD) group
  Interventions: Other: Hysteroscopy

INTERVENTIONS:
Other: Hysteroscopy — 1. Three groups of patients will be enrolled: Natural labour group, Cesarean scar group and Cesarean with diverticulum (PCSD) group;
  2. Hysteroscopy will be carried out for uterine cavity examine and the specimen collection for further microflora analysis and inflammation marker detection;
  3. ART will be carried out with standard protocol and the clinical outcome will be recorded;
  4. The primary outcome of the study is the comparation of species and communities of uterine microflora and inflammatory markers of the female uterus among three groups. The secondary outcome is biochemical pregnancy rate, clinical pregnancy rate, embryo implantation rate and live birth rate.
  Other Names: assisted reproductive medicine

SUMMARY:
Mode of delivery affects the success rate of assisted reproductive techniques (ART). In this case study, the investigators will evaluate changes in the bacterial ecology and inflammatory markers of the female uterus with different delivery modes. We will investigate whether the dominate endometrial microflora is interrupted by the Cesarean section in the infertile women undergoing ART, and the potential mechanism will also be further explored prospectively.

DETAILED DESCRIPTION:
The highly prevalence of cesarean section rate in China had drawn great attention world widely. Post-cesarean section scar diverticulum ( PCSD) is a poor healing of the local incision after Cesarean section which happened in19.4%~88% of patients. The cavity is formed by the original incision connected with the uterine cavity. Patients with diverticulum are often accompanied by prolonged menstruation and uterine effusion, which may accompany with endometrial inflammation and impair embryo implantation rate.

Though Cesarean section plays an important role in the treatment of dystocia and also decreasing perinatal mortality, it may impact natural conception and the success rate of ART in secondary infertile patients. Data from other researchers have revealed that Cesarean scar may related to poor pregnancy outcome during ART treatment. We have retrospectively analyzed the pregnancy outcome of ART treatment in patients who have had live birth previously from January 2014 to May 2018. The biochemical pregnancy rate, embryo implantation rate and clinical pregnancy rate are all lower in patients with Caesarean section compared to patients after natural labour, the clinical data is even worse in patients with PCSD. The results suggest a close correlation between the outcome of assisted reproductive therapy and the uterine condition. Further evaluations are required related to whether the dominate endometrial microflora is interrupted by the Cesarean section in the infertile women undergoing ART, and the potential mechanism will also be explored accordingly. A single-center, prospective, case-control study will be carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Women age ≥20 years and ≤40 years.
2. infertile Women with previously live birth.
3. Previous failed transfer cycle ≤2
4. Didn't participate in other clinical subjects within three months.
5. Written informed consent.

Exclusion Criteria:

1. surgery history including: Ovariectomy, myomectomy, adenomyomectomy.
2. Uterine diseases including: uterine malformation, submucosal uterine fibroids and intrauterine adhesion.
3. One of couple has abnormal karyotype.
4. Recurrent abortion ≥2.
5. Untreated hydrosalpinx.
6. History of tuberculosis (pulmonary tuberculosis, pelvic tuberculosis etc.).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile patients who had live birth previously and met the criteria, required for IVF treatment from Aug 2019 to Aug 2022 in our center.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Species and communities of uterine microflora | 1-2 year
  Use the swab to scrape endometrium. Characterization of species and communities of uterine microflora will use bacterial DNA microarray analysis. Normally, the uterine cavity used to being thought a sterile space.
Inflammatory markers of the female uterus | 1-2 year
  Use the swab to scrape endometrium. Characterization of inflammatory markers of the female uterus will use human cytokines measuring. The cytokines will include IL2,IL4,SDF-1α , etc. Use the natural labor group as control group, and see differentiation among the three group.

SECONDARY OUTCOMES:
Clinical pregnancy rate | 1-2 year
  Clinical pregnancy means pregnancy sac is seen intrauterine under ultrasound 7 weeks after embryo transferred.
  Clinical pregnancy rate(%): number of clinical pregnancy/transferred cycle.
Biochemical pregnancy rate | 1-2 year
  Biochemical pregnancy rate(%): number of biochemical pregnancy/transferred cycle.
Embryo implantation rate | 1-2 year
  Embryo implantation rate(%): number of gestational sac / transferred embryo.
Live birth rate | 1-2 year
  Live birth rate(%): number of live birth/ transferred cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Yang, M.D. & Ph.D, Study Chair — The Sixth Affiliated Hospital, Sun Yat-sen University; Xaoyan Liang, M.D. & Ph.D, Study Director — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital,Sun Yat-Sen University, Guandong, China